CLINICAL TRIAL: NCT01087801
Title: A Placebo Controlled, Double-Blind, Parallel, Multicenter Study of Synthetic Human Secretin (ChiRhoStim®) Administered Intravenously to Stimulate Exocrine Pancreas Fluid Secretion for Collection Via Endoscope and Laboratory Analysis of DNA Markers
Brief Title: A Study of Synthetic Human Secretin (ChiRhoStim®) Administered Intravenously to Stimulate Exocrine Pancreas Fluid Secretion for Collection Via Endoscope and Laboratory Analysis of DNA Markers
Acronym: CRC2006-05
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ChiRhoClin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2006-05
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Pancreatic Disease
Keywords: Genetic End Marker
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChiRhoStim (Active Comparator): Human Secretin for Injection
  Interventions: Drug: ChiRhoStim
- Placebo (Placebo Comparator): Saline for Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ChiRhoStim — Human Secretin for Injection
  Arms: ChiRhoStim
Drug: Placebo — Saline for Injection
  Arms: Placebo

SUMMARY:
The following are the study hypothesis:

* Secretin administration compared to placebo will result in a statistically significantly greater percentage of collected fluid samples being predominantly of exocrine pancreas origin when samples are duodenal aspirates.
* Secretin administration compared to placebo will result in a statistically significantly greater percentage of collected fluid samples meeting the minimum specifications for use in the indicated laboratory test of DNA mutational analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Documented or suspected diagnosis of chronic pancreatitis or suspected diagnosis of pancreatic cancer.
2. Undergoing Endoscopic Procedure.
3. Age ≥ 18 years.
4. Willing and able to sign informed consent, meeting IRB guidelines.
5. Willing and able to meet all study requirements and obligations.

Exclusion Criteria:

1. Ongoing, active pancreatitis at the time of the procedure.
2. Known adverse reaction to secretin.
3. Recent (within one month) use of medication that can potentially cause pancreatitis, such as metronidazole, tetracycline, sulfonamides.
4. Use of anticholinergic medication within 7 days of study.
5. Pregnant women, nursing mothers, or women of childbearing potential not employing appropriate contraception. Acceptable methods of birth control are: intrauterine device, implantable progesterone device, progesterone intramuscular injection, oral contraceptive (started at least one month prior to Visit 1 and continuing for the duration of the trial), contraceptive patch, condoms with spermicide or abstinence.
6. Any medical condition which in the judgment of the Principal Investigator makes participation of the patient in the study medically unwarranted.
7. Known complete obstruction of the pancreatic duct.
8. Patients who have received an investigational product/drug or device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Burton, M.D., Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ChiRhoStim: Human Secretin for Injection 0.1 mL/kg IV
- Placebo: Saline for Injection 0.1 mL/kg IV
Period: Overall Study
Arm/Group | ChiRhoStim | Placebo
Started | 30 | 34
Completed | 26 | 29
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChiRhoStim | Placebo | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants] — The demographic data represents the intent to treat group when data was provided in cases where no demographic data was provided for a parameter, the number of observations was correspondenly reduced.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 23 | 27 | 50
    >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 49.6 (15.5) | 47.2 (12.3) | 48.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Sample
Description: Is Volume ≥ 3.5 mL Is HCO3 concentration ≥ 40 mEq/L Is DNA mutational analysis (K-ras-2 gene Fluorescence peak height ≥ 50 Relative Florescence Units panel assessable markers informative ≥ 8).
  (Note- The outcome value is boolean (yes or no) as an answer).
Time Frame: First 5 minutes after treatment administration
Reporting Status: Not Posted

2. Primary Outcome: Volume of Fluid ≥ 3.5mL (Boolean Expression Evaluated as Yes or no).
Description: Volume of pancreatic fluid. The volume is the number of mL of pancreatic fluid.
Time Frame: First 5 minutes after treatment administration
Measure: Number; unit: Participants
Arm/Group | ChiRhoStim | Placebo
Number analyzed (Participants) | 26 | 29
Participants
  Yes | 25 | 2
  No | 1 | 27

ADVERSE EVENTS:
Arm/Group | ChiRhoStim | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/34
Other Adverse Events (participants affected / at risk) | 0/30 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No